CLINICAL TRIAL: NCT06374459
Title: A Phase Ib/II Trial of Zunsemetinib in Combination With Capecitabine in Patients With Hormone Receptor-Positive and HER2-Negative Metastatic Breast Cancer With Bone Metastasis
Brief Title: Zunsemetinib in Combination With Capecitabine in Patients With Hormone Receptor-Positive and HER2-Negative Metastatic Breast Cancer With Bone Metastasis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202406065; BC200714 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-04-10; First posted 2024-04-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hormone Receptor Positive HER-2 Negative Metastatic Breast Cancer
Keywords: Zunsemetinib; ATI-450; MK-2; Bone metastasis; Breast Cancer; HR-positive/HER2-negative; Capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Zoledronic Acid; Denosumab

STUDY DESIGN:
Intervention Model Description: The Phase I portion of the study is sequential and patients will not be randomized and the Phase II portion is parallel and patients will be randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase Ib: Zunsemetinib + Capecitabine (Experimental): Patients will receive zunsemetinib by mouth (PO) twice per day (BID) at an assigned dose along with capecitabine (1000 mg/m^2 PO BID on Days 1-14 an every 21-day cycle). For patients enrolled in phase Ib, capecitabine is dosed on days 2-15 during cycles 1-2. Dose escalation of zunsemetinib will utilize a 3+3 design. A maximum of 3 dose levels of zunsemetinib will be tested, and the two highest dose levels which did not lead to more than 1 of 6 patients with DLT in cycle 1 will be chosen as the RP2D-L1 and RP2D-L2 for Phase II. If only one dose level of zunsemetinib was found tolerable, then only one RP2D will be chosen for Phase II.
  Interventions: Drug: Zumsemetinib; Drug: Capecitabine
- Phase II Arm 1: Standard of care anti-resorptive + Capecitabine (Active Comparator): Standard of care anti-resorptives will consist of bisphosphonate (zoledronic acid) is to be administered every 4-12 weeks, or denosumab is to be administered every 4-6 weeks, as per physician choice and institutional practice. In general, capecitabine will be taken twice daily at a dose of 1000 mg/m^2 on Days 1 through 14 of every 21-day cycle. The first 4 patients enrolling to phase II will take capecitabine on a different schedule for PK purposes in Cycles 1 and 2 ONLY. Patients will take capecitabine at a dose of 1000mg/m^2 on Days 2 through 15 of Cycles 1 and 2, and then on Days 1 through 14 starting with Cycle 3.
  Interventions: Drug: Capecitabine; Drug: Zoledronic acid; Drug: Denosumab
- Phase II Arm 2: Zunsemetinib (RP2D-L1) + Capecitabine (Experimental): Patients will receive zunsemetinib by mouth (PO) twice per day (BID) at an assigned dose. In general, capecitabine will be taken twice daily at a dose of 1000 mg/m^2 on Days 1 through 14 of every 21-day cycle. The first 4 patients enrolling to phase II will take capecitabine on a different schedule for PK purposes in Cycles 1 and 2 ONLY. Patients will take capecitabine at a dose of 1000mg/m^2 on Days 2 through 15 of Cycles 1 and 2, and then on Days 1 through 14 starting with Cycle 3.
  Interventions: Drug: Zumsemetinib; Drug: Capecitabine
- Phase II Arm 3: Zunsemetinib (RP2D-L2) + Capecitabine (Experimental): Patients will receive zunsemetinib by mouth (PO) twice per day (BID) at an assigned dose. In general, capecitabine will be taken twice daily at a dose of 1000 mg/m^2 on Days 1 through 14 of every 21-day cycle. The first 4 patients enrolling to phase II will take capecitabine on a different schedule for PK purposes in Cycles 1 and 2 ONLY. Patients will take capecitabine at a dose of 1000mg/m^2 on Days 2 through 15 of Cycles 1 and 2, and then on Days 1 through 14 starting with Cycle 3. If only one dose level of zunsemetinib plus capecitabine was found tolerable in phase Ib testing, the phase II trial will proceed with 2:1 two-arm randomization with Arm 2 of capecitabine plus zunsemetinib and Arm 1 of capecitabine plus standard of care anti-resorptive agent.
  Interventions: Drug: Zumsemetinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Zumsemetinib — Patients should take zunsemetinib at approximately the same times every day, with or without food with 8 oz of water.
  Other Names: ATI-450
  Arms: Phase II Arm 2: Zunsemetinib (RP2D-L1) + Capecitabine; Phase II Arm 3: Zunsemetinib (RP2D-L2) + Capecitabine; Phase Ib: Zunsemetinib + Capecitabine
Drug: Capecitabine — Patients should take capecitabine at approximately the same times every day, within 30 minutes after a meal.
Drug: Zoledronic acid — Standard of care. Will receive zoledronic acid or denosumab.
  Arms: Phase II Arm 1: Standard of care anti-resorptive + Capecitabine
Drug: Denosumab — Standard of care. Will receive zoledronic acid or denosumab.
  Arms: Phase II Arm 1: Standard of care anti-resorptive + Capecitabine

SUMMARY:
This is a phase Ib/II study evaluating the safety and efficacy of zunsemetinib (ATI-450) with capecitabine in patients with hormone receptor-positive and HER2-negative (HR+/HER2-) metastatic breast cancer (MBC).

ELIGIBILITY:
Inclusion Criteria for both Phase Ib and Phase II:

* Hormone receptor-positive, HER2-negative metastatic breast cancer.
* Measurable or non-measurable but evaluable disease by RECIST v1.1.
* Candidate for capecitabine treatment per physician decision. See below phase-specific eligibility criteria for further guidance.
* No more than one prior chemotherapy for metastatic disease.
* Patient must have received prior endocrine therapy with CDK4/6 inhibitor.
* If patient is on denosumab or zoledronic acid prior to enrollment, patient must have been on the regimen for at least 6 months prior to study. However, a washout of 3 weeks is required prior to C1D1.
* At least 18 years of age.
* ECOG performance status 0, 1, or 2
* Life expectancy of at least 12 weeks.
* Adequate bone marrow and organ function as defined below:

  * Leukocytes ≥ 3 K/cumm
  * Absolute neutrophil count (ANC) ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Total bilirubin ≤ 1.5 x IULN (or total bilirubin ≤ 3 mg/dL if patient has known Gilbert Syndrome)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance > 60 mL/min by Cockcroft-Gault
  * Calcium within normal limits
* Women of childbearing potential and men who are heterosexually active must agree to use adequate contraception as specified in the protocol. Contraception should continue for 6 months (for women) or 3 months (for men) after the end of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.
* Patients must have archival tissue sample available from prior metastatic biopsy. If no tissue is available, patient may still be able to enroll with PI approval.

Inclusion Criteria for both Phase Ib:

* Presence of bone metastasis is not required.
* Candidate for, or currently on stable doses of capecitabine, defined as capecitabine: 1000 mg/m^2 BID, 14 days on and 7 days off. A stable dose of capecitabine is defined as no more than grade 1 AEs related to capecitabine on the 1000 mg/m^2 BID, 14 days on and 7 days off dose for at least 1 cycle. Capecitabine is not counted as a prior chemotherapy regimen in these patients.

Inclusion Criteria for Phase II:

* Progressive bone metastasis per the most recent tumor imaging studies by RECIST 1.1 or clinical progression (such as worsening bone pain, elevation of tumor marker) per treating physician.

Exclusion Criteria for both Phase Ib and Phase II:

* Patients may not have received the following investigational or SOC therapies within the below specified time frames prior to C1D1:

  * Radiation therapy within 1 week
  * Systemic chemotherapy, including antibody drug conjugates with chemotherapy payload, within 3 weeks.
  * Immunotherapy within 3 weeks
  * Oral chemotherapy or molecularly targeted therapy within 5 half-lives of the agent.
  * Endocrine therapies do not have a required washout and may be continued until C1D1.
  * Strong and moderate CYP3A4 and CYP2C8 inhibitors (including grapefruit), strong and moderate CYP3A and CYP2C8 inducers, and drugs with QT prolonging potential within 5 half-lives of the agent.
* Untreated brain metastases. Patients with treated brain metastases are eligible if they show no evidence of progression and are off steroids.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to zunsemetinib or other agents used in the study.
* History of acute, untreated skeletal related events (SRE) or active untreated SRE or a change or an anticipated change in the SOC anti-resorptive agents after entering the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of C1D1.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to Cycle 1 Day 1. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.
* Screening resting QTcF above 470 msec.

Exclusion Criteria for Phase Ib:

* Capecitabine within 2 weeks prior to C1D1. Patients may be currently taking capecitabine, but must not have dosed within 2 weeks prior to C1D1 for study correlative purposes.

Exclusion Criteria for Phase II:

* Prior capecitabine in the metastatic setting.
* History of other malignancy, unless all treatment was completed and patient had no evidence of disease within 2 years of C1D1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2032-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (Phase Ib only) | From start of treatment through 30 days after end of treatment (estimated to be 11 months)
Recommended phase II dose of zunsemetinib (Phase Ib only) | Through end of 1st cycle (each cycle is 21 days)
Number of participants with dose-limiting toxicities (Phase Ib only) | Through end of 1st cycle (each cycle is 21 days)
Percent change in serum CTX (Phase II only) | Baseline and Day 1 of week 7
Progression-free survival (PFS) (Phase II only) | From start of treatment through completion of follow-up (estimated to be 3 years and 10 months)

SECONDARY OUTCOMES:
Treatment-induced changes in DEXA BMD (g/cm^2) at hip and spine (Phase Ib only) | Baseline, end of cycle 8 (each cycle is 21 days), and end of treatment (estimated to be 10 months)
Treatment-induced changes in sCTX by clinical assay (Phase II only) | Baseline, cycle 1 day 1 pre-dose, cycle 1 day 8 pre-dose, cycle 1 day 15 pre-dose, day 1 of subsequent cycles (each cycle is 21 days), and end of treatment (estimated to be 10 months)
Objective response rate (ORR) (Phase II only) | Through completion of treatment (estimated to be 10 months)
Clinical benefit rate (Phase II only) | Through completion of treatment (estimated to be 10 months)
Overall survival (OS) (Phase II only) | From start of treatment through completion of follow-up (estimated to be 3 years and 10 months)
Treatment-induced changes in DEXA BMD (g/cm^2) at hip and spine (Phase II only) | Baseline, end of cycle 8, and end of treatment (estimated to be 10 months)
Treatment-induced changes in quality of life as measured by EORTC QLQ-C30 (Phase II only) | Prior to start of 1st treatment, cycle 5 day 1, every 4 cycles thereafter (each cycle is 21 days), and at the time of progression (estimated to be 3 years and 10 months)
Treatment-induced changes in pain as measured by Brief Pain Inventory (BPI) (Phase II only) | Prior to start of 1st treatment, cycle 5 day 1, every 4 cycles thereafter (each cycle is 21 days), and at the time of progression (estimated to be 3 years and 10 months)
Number of participants with adverse events (Phase II only) | From start of treatment through 30 days after end of treatment (estimated to be 11 months)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia X Ma, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
The investigator will share deidentified individual patient level data upon request after publication of the trial results.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of trial results.
Access Criteria: Data use agreement will be needed and contact can be made with the Principal Investigator for requests.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu